CLINICAL TRIAL: NCT06926712
Title: The Effect of Vitamin E Supplementation on Hospital Stay Duration in Non-cyanotic Heart Disease Children With Lower Respiratory Tract Infections - Randomized Controlled Trial
Brief Title: The Effect of Vitamin E Supplementation on Hospital Stay Duration in Non-cyanotic Heart Disease Children With Lower Respiratory Tract Infections
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Ahmed Mohamed, Safaa Ahmed Mohamed Ali, lecturer assesstant at family medicine department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: safaa1451995protocol
Record Dates: First submitted 2025-03-12; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Disease
Keywords: RTI-VIT E- CHD
MeSH Terms: conditions — Respiration Disorders | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Active Comparator): The intervention group will receive vitamin E in an appropriate dose during the hospital stay with the treatment protocol for chest infection
  Interventions: Drug: Vitamin E
- control group (No Intervention): The control group will receive the treatment protocol for chest infection only or with placebo instead of vitamin E.

INTERVENTIONS:
Drug: Vitamin E — dose of vitamin E in an appropriate dose for age during hospital stay for intervention group
  Arms: intervention

SUMMARY:
Congenital heart disease can lead to serious health issues, particularly an increased risk of infections, specifically respiratory infections. Lower respiratory tract infections are the fifth leading cause of death globally. Also considered a significant cause of morbidity and mortality among children with congenital heart disease.

In Egypt, it is estimated that 10% of deaths in children under the age of 5 years are probably caused by lower respiratory tract infections and other acute respiratory infections. common non-cyanotic CHD like Ventricular septal defect predispose to bronchopneumonia.

Hemodynamically significant congenital heart disease with pulmonary congestion increases the risk of lower respiratory tract infections and hospitalizations. This relies on several modifiable risk factors, including low socioeconomic status, poor diet, overcrowding, prematurity, male gender, and exposure to secondhand smoke.

Micronutrients play a crucial role in strengthening the immune system. Many Studies have shown that when children are supplemented with various micronutrients, they experience fewer episodes of acute respiratory infections, and the duration and severity of these infections are reduced.

Vitamin E is essential for immune system function and may lower disease risk by enhancing immune responses. It protects neurons and respiratory mucosa from oxidative damage and has been linked to a reduced incidence of asthma and inflammation, potentially safeguarding young children from atopy and wheezing.

There are no available studies in our locality about the effect of vitamin E supplementation on the length of hospital stay for non-cyanotic cardiac patients with lower respiratory tract infections.

DETAILED DESCRIPTION:
Congenital heart disease can lead to serious health issues, particularly an increased risk of infections, specifically respiratory infections. Lower respiratory tract infections are the fifth leading cause of death globally. Also considered a significant cause of morbidity and mortality among children with congenital heart disease.

In Egypt, it is estimated that 10% of deaths in children under the age of 5 years are probably caused by lower respiratory tract infections and other acute respiratory infections. common non-cyanotic CHD like Ventricular septal defect predispose to bronchopneumonia.

Hemodynamically significant congenital heart disease with pulmonary congestion increases the risk of lower respiratory tract infections and hospitalizations. This relies on several modifiable risk factors, including low socioeconomic status, poor diet, overcrowding, prematurity, male gender, and exposure to secondhand smoke.

Micronutrients play a crucial role in strengthening the immune system. Many Studies have shown that when children are supplemented with various micronutrients, they experience fewer episodes of acute respiratory infections, and the duration and severity of these infections are reduced.

Vitamin E is essential for immune system function and may lower disease risk by enhancing immune responses. It protects neurons and respiratory mucosa from oxidative damage and has been linked to a reduced incidence of asthma and inflammation, potentially safeguarding young children from atopy and wheezing.

There are no available studies in our locality about the effect of vitamin E supplementation on the length of hospital stay for non-cyanotic cardiac patients with lower respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients are diagnosed with non-cyanotic heart disease associated with severe lower respiratory tract infection. ⁃ The patients are aged 2 months to 5 years of both sexes.

Exclusion Criteria:

* Pediatric patients that have other congenital anomalies other than CHD.

  * Those with chronic respiratory diseases such as asthma, bronchiectasis, etc.).
  * Immunocompromised patients, such as those who receive steroids or chemotherapy, etc.
  * Pediatric patient that received vitamin E in the previous month.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
the length of hospital stay | During the intervention
  The effect of vitamin E supplementation on the length of hospital stay in non-cyanotic cardiac pediatric patients with lower respiratory tract infections.

SECONDARY OUTCOMES:
risk factors | During the intervention
  To assess the impact of identified risk factors (e.g., prematurity, malnutrition, severity of pneumonia, and different age groups) on hospital length of stay.
  - To determine the incidence of complications (e.g., need for ICU, mechanical ventilation, congestive heart failure) concerning identified risk factors.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] [1] M. M. Djer and D. B. S. , Emilda Osmardin, Badriul Hegar, "Increased Risk of Recurrent Acute Respiratory Infections in Children with Congenital Heart Disease: A Prospective Cohort Study," Indones. Biomed. J., vol. 12, no. 4, p. p.288-389, 2020, doi: 10.18585/inabj.v12i4.1262. [2] E. Kılıçoğlu and Z. Ü. Tutar, "Evaluation of Children with Congenital Heart Disease Hospitalized with the Diagnosis of Lower Respiratory Tract Infection," J. Pediatr. Res., vol. 5, no. July 2017, pp. 32-36, 2018. [3] Z. Chen, "Circulating micronutrient levels and respiratory infection susceptibility and severity : a bidirectional Mendelian randomization analysis," no. August, 2024, doi: 10.3389/fnut.2024.1373179. [4] A. M. M. Hamed, Y. T. Kassem, H. K. Fayed, and A. M. Solaiman, "Serum zinc levels in hospitalized children with pneumonia: a hospital-based case-control study," Egypt. J. Bronchol., vol. 13, no. 5, pp. 730-737, 2019, doi: 10.4103/ejb.ejb_30_19. [5] N. K. Jat, D. K. Bhagwani, N. Bhutani, U. Sharma, R. Sharma, and R. Gupta, "Assessment of the prevalence of congenital heart disease in children with pneumonia in tertiary care hospital : A cross-sectional study," Ann. Med. Surg., vol. 73, no. November 2021, p. 103111, 2022, doi: 10.1016/j.amsu.2021.103111. [6] O. Investigation, "The Role of the Micronutrients; Vitamin A, Vitamin B12, Iron, Zinc, Copper Levels of Children with Lower Respiratory Tract Infections," pp. 105-109, 2005, doi: 10.5152/ced.2014.1319. [7] M. X. Wang, J. Koh, and J. Pang, "Association between micronutrient deficiency and acute respiratory infections in healthy adults : a systematic review of observational studies," pp. 1-12, 2019. [8] P. C. Calder and P. Yaqoob, "Nutrient Regulation of the Immune Response," Present Knowl. Nutr. Tenth Ed., no. January, pp. 688-708, 2012, doi: 10.1002/9781119946045.ch44. [9] S. Wu and A. Wang, "Serum level and clinical significance of vitamin E in pregnant women with allergic rhinitis," J. Chinese Med. Assoc., vol. 85, no. 5, pp. 597-602, 2022, doi: 10.1097/JCMA.0000000000000723. [10] S. I. Fahmy, L. M. Nofal, S. F. Shehata, H. M. El, and H. K. Ibrahim, "Updating indicators for scaling the socioeconomic level of families for health research," pp. 1-7, 2015, doi: 10.1097/01.EPX.0000461924.05829.93. [11] J. Thokngaen and W. Karoonboonyanan, "Pediatric respiratory severity score evaluates disease severity of respiratory tract infection in children," Chulalongkorn Med. J., vol. 63, no. 1, pp. 41-46, 2019, doi: 10.14456/clmj.1476.6. [12] T. Bohn et al., "Scientific opinion on the tolerable upper intake level for vitamin E," vol. 22, pp. 1-104, 2024, doi: 10.2903/j.efsa.2024.8953.